CLINICAL TRIAL: NCT05758428
Title: A Phase 1, Open-Label, Single and Multiple Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Nebulized Ensifentrine in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Nebulized Ensifentrine in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuance Pharma (shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPL554-AHC001
Record Dates: First submitted 2023-02-14; First posted 2023-03-07 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Subjects will receive a 3 mg ensifentrine single dose, followed by 3 mg repeated dose (twice daily, BID).
  Interventions: Drug: Ensifentrine
- Cohort 2 (Experimental): Subjects will receive two single doses of 1.5 mg and 6 mg ensifentrine, separated by at least a 7-day washout period using crossover design.
  Interventions: Drug: Ensifentrine

INTERVENTIONS:
Drug: Ensifentrine — 14 Subjects enrolled will use one 3 mg/2.5 mL ampule for the 3 mg dose, subjects will receive a 3 mg ensifentrine single dose, followed by 3 mg repeated dose (twice daily, BID). On the dosing day (Day 1), subjects will receive a single dose of 3 mg ensifentrine. On Day 4, subjects will receive multiple doses of 3 mg ensifentrine BID for 3 days (Day 4 to Day 6), and a morning dose will be administered on Day 7.
  Arms: Cohort 1
Drug: Ensifentrine — 14 subjects will be enrolled in this cohort, then randomly assigned to one of 2 treatment sequences (6mg and 1.5mg single dose). Subjects will 2 different dose levels of study drug. Two 3 mg/2.5 mL ampules will be needed for the 6 mg dose (5 mL total volume) and the 1.5 mg dose will be achieved using an appropriate dilution protocol described in the pharmacy manual.
  Other Names: Placebo
  Arms: Cohort 2

SUMMARY:
This is a phase 1, open-label, parallel cohort study to evaluate the PK, safety and tolerability of nebulized ensifentrine following administration of single and multiple doses in healthy Chinese male subjects.

DETAILED DESCRIPTION:
This study consists of two cohorts, and approximately a total of up to 28 healthy male subjects, 14 subjects in Cohort 1, and 14 subjects in Cohort 2, will be enrolled. Cohort 2 will be randomly assigned to Sequence 1 and Sequence 2 according to the ratio of 1:1.

Treatment Group

1. Cohort 1: subjects will receive a 3 mg ensifentrine single dose, followed by 3 mg repeated dose (twice daily, BID).
2. Cohort 2: subjects will receive two single doses of 1.5 mg and 6 mg ensifentrine, separated by at least a 7-day washout period using crossover design.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (18-50 yrs) who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECG without abnormality or with abnormality of no clinical significance;
2. A male subject must agree to use contraception as detailed in the protocol from the screening visit to within 30 days of the last dose after study completion and refrain from donating sperm during this period;
3. Subjects never smoke or is ex-smoker for ≥ 12 months,never chewing tobacco within 90 days prior to screening;
4. 3. Body weight must be ≥ 50 kg and body mass index (BMI) between 18.0 and 30.0 kg/m2.

Exclusion Criteria:

1. History or current malignancy of any organ system, treated or untreated within the past 5 years;
2. Known allergy, immune reaction, or intolerance to ensifentrine or any of the excipients of the formulation and/or ineligible to receive ensifentrine;
3. Subjects with the history of pulmonary and cardiovascular disease;
4. Any chronic condition or disease, including but not limited to: Metabolism, endocrine (such as diabetes, hypothyroidism/hyperthyroidism), liver, kidney, gastrointestinal tract, hematology or nervous system and other diseases;
5. Respiratory tract infection (upper and/or lower) treated with antibiotics within 12 weeks of screening visit;
6. Current infection of clinical significance or known ongoing inflammatory condition;
7. Live or attenuated vaccine(s) within 1 month prior to screening, or plan to receive such vaccines during the study;
8. Immunotherapy within 30 days of screening;
9. Subjects who participated in any other interventional clinical trials within 3 months prior to screening;
10. Subjects who have used any drugs that inhibit or induce liver metabolism of drugs within 30 days prior to screening or have used any drugs within 14 days prior to screening;
11. Subjects who have a history of alcohol or drug abuse, or have used any drug abuse within 6 months before screening;
12. Subjects with a positive alcohol breath test, or a positive urinalysis screening test or a positive smoke test;
13. Creatinine clearance < 80mL/min by Cockcroft-Gault formula;
14. Subjects who have clinically significant abnormalities in physical examination, vital signs, chest x-ray, and laboratory examinations;
15. Pulmonary function test: Subjects who have measured value of forced expiratory volume in first second (FEV1) / predicted value of FEV1 ≤ 80% or forced vital capacity (FVC) ≤ 80% of predicted value or any other clinically significant abnormality;
16. Subjects who have any of abnormal findings in 12-lead ECG or any other clinically significant abnormality;
17. Subjects who have undergone surgery within 6 months prior to the dosing of the study drug or who have undergone surgery within 4 weeks prior to the dosing of the study drug or who plan to undergo surgery during the trial;
18. Donated blood or blood products or had substantial loss of blood (more than 300 mL) within 56 days prior to the first administration of study treatment.
19. Unwilling to follow the lifestyle considerations;
20. Any other reason that the investigator considers the patient unsuitable to participate in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Cmax of RPL554 | 0 to 72 hours
  Blood PK sampling for RPL554 concentration
AUC0-t of RPL554 | 0 to 72 hours
  Area under the plasma concentration from time 0 to the last collection time after drug administration
Tmax of RPL554 | 0 to 72 hours
  Time to maximum observed plasma concentration
t1/2 of RPL554 | 0 to 72 hours
  Half-life of RPL554

SECONDARY OUTCOMES:
Adverse events | From the first dose usage to the end of the study, approxiamtely up to 15 days
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No